CLINICAL TRIAL: NCT00298480
Title: Dynamic Cervical Change: Prediction of Preterm Labor in Symptomatic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Memorial Health Services Research Council (Other)
Other Study IDs: 230-04s
Record Dates: First submitted 2006-03-01; First posted 2006-03-02 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Dynamic Cervical Change in Preterm Labor Patients
Keywords: preterm labor; transvaginal ultrasound; dynamic cervical change
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Transvaginal ultrasound of the cervix has become a common tool to evaluate patients who are at risk for preterm delivery. A shortened cervical length has been associated with an increased risk of preterm delivery. Dynamic cervical change is visible shortening(>6mm) of the cervix seen during the ultrasound examination. Prior studies have shown that the presence of dynamic change in patients with a shortened cervical length(<3cm) is not independently predictive of preterm delivery. However, a subset of patients with normal initial cervical length(>3cm) and dynamic change did demonstrate an increased rate of preterm delivery. Because this was a small sub-group, the present study was designed to obtain a larger sample size for further evaluation. The second focus of this study involves patients with a dilated cervix and whether cervical length adds predictive value to gestational age at delivery.

Patients presenting to with symptomatic preterm labor(vaginal pressure or uterine contractions), who consent to the study, will undergo the standard evaluation for preterm labor(described in detail below.) The only additional evaluation is a prolonged transvaginal ultrasound of approximately 10 minutes to evaluate for the presence of dynamic change during a contraction.

Null hypothesis:

Symptomatic preterm labor patients, with normal initial cervical length(>3cm), who exhibit dynamic cervical change deliver at a gestational age equal to those without dynamic change.

Alternative hypothesis:

Symptomatic preterm labor patients, with normal initial cervical length(>3cm), who exhibit dynamic cervical change deliver at an earlier gestational age than those without dynamic change.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the ages of 18 and 45 years.
* Intrauterine pregnancy with gestational age between 22 0/7 and 34 6/7 weeks gestation.
* Presenting with symptomatic preterm labor (e.g. Regular uterine contractions, uterine cramping, or pelvic pressure).

Exclusion Criteria:

* Cervical cerclage
* Ruptured membranes noted on initial speculum examination
* Cervical os dilation >4 cm noted on initial digital examination
* Known HIV-positive or active HSV(to minimize the risk of perinatal exposure)
* Presence of multiple genital warts
* Patients under extreme duress from their uterine contractions

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Enrollment: 220
Dates: Start 2005-02; Study Completion 2007-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte A Clock, M.D., Principal Investigator — University of California, Irvine; James Kurtzman, M.D., Principal Investigator — University of California, Irvine
Locations (3):
- United States (3):
  - Saddleback Memorial Medical Center, Laguna Hills, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - University of California, Irvine Medical Center, Orange, California